CLINICAL TRIAL: NCT02694692
Title: Trial of Repeated Analgesia With Kangaroo Care - 18 Month Follow-up
Acronym: TRAKC18
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IWK Health Centre (Other)
Collaborators: Nova Scotia Health Research Foundation (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1017737
Record Dates: First submitted 2016-02-24; First posted 2016-02-29 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Pain; Development
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Follow-up: No further interventions are planned for this trial and the three pain management interventions from the original study (NCT01561457) will remain our comparison groups (Kangaroo Mother Care alone, Sucrose alone, and Kangaroo Mother Care & Sucrose). All participants will be invited to back to the IWK Health Centre to receive their Vaccinations at 2, 6, 12 and 18 month time points as well as for their Neurodevelopment assessment at 18 corrected age (BSID-III).
  Interventions: Procedure: Vaccinations at 2, 6, 12 and 18 month; Behavioral: Neurodevelopment assessment at 18 corrected age

INTERVENTIONS:
Procedure: Vaccinations at 2, 6, 12 and 18 month — Participants will be invited back to IWK Health Centre at time points that correspond to their 2, 6, 12 and 18 month vaccinations and will receive their vaccinations according to Nova Scotia schedule.
Behavioral: Neurodevelopment assessment at 18 corrected age — During the 18 month follow-up visit, the infants will also undergo neurodevelopmental assessment. Trained medical assessors also blind to original study group assignment will examine the child using the BSID-III Cognitive and Motor Sections. Participants will also be contacted at the infants 18 month corrected postnatal age for the BSIDIII. Parents will be asked to complete the Early Childhood Behaviour Questionnaire and the Brief Infant Toddler Social Emotional Assessment.

SUMMARY:
The primary aim for this study is to determine if maternal Kangaroo Care (KC) provided during painful procedures in early life will mitigate stress release and will improve neurobehavioural outcomes in infants, decrease subsequent pain response, and enhance maternal-child interaction beyond the period of hospitalization.

DETAILED DESCRIPTION:
Background: Infants in the Neonatal Intensive Care Unit receive an average of 7 painful procedures daily yet less than half receive interventions to manage pain. Importantly, there are adverse long-term effects associated with untreated pain. Moreover, the developmental trajectory of an infant born preterm is further compromised by prolonged periods of separation from their mothers during their hospital stay that also impacts mother-infant relationships. Thus, there is a crucial need to minimize procedural pain and associated consequences. Kangaroo Care (KC) is an effective strategy for reducing procedural pain and promoting mother-infant interactions in infants demonstrated in multiple clinical trials and systematic reviews. Not known is the impact of consistent KC for pain on long term outcomes. The primary aim for this study is to determine if maternal KC provided during painful procedures in early life will mitigate stress release and will improve neurobehavioural outcomes in infants, decrease subsequent pain response, and enhance maternal-child interaction beyond the period of hospitalization.

Research Design: Using a randomized clinical trial follow up design, mother-infant dyads taking part in the current CIHR and NSHRF-funded TRAKC trial (randomized to one of three interventions during all routine clinically necessary painful procedures for the duration of their initial neonatal intensive care unit hospital stay (KC/placebo; sucrose alone, considered to be standard care; or KC/ sucrose) will be compared on neurobehavioural outcomes up to 18 months.

Procedure: Eligible mother-infant dyads will be contacted prior to routine 2, 6, 12 and 18 month clinic visits where during these visits, infants will undergo an immunization and naturalistic observations will be recorded. Coders blinded to the study will score pain intensity and maternal comforting behavior using validated measures. At the 18 month visit, trained medical assessors blind to group assignment will perform the primary outcome measure, Bayley Scales of Infant Development (3rd ed) (BSID-III).

Outcomes: The investigators hypothesize that infants from the current TRAKC trial who were assigned to either KC group (alone or in combination with sucrose) when compared to those infants in the sucrose alone group will have: Primary outcome: H1. higher scores on the BSID-III at 18 months corrected postnatal age. Secondary outcomes: H2. higher scores in socio-affective development (Social-Emotional axis of the BSID-III and the Brief Infant Toddler Social Emotional Assessment (BITSEA); H3. lower scores on Negative Affectivity, higher scores on Surgency/Extraversion and Effortful Control as measured by the Early Childhood Behavior Questionnaire (ECBQ); H4. lower pain scores measured using the Modified Behavioral Pain Scale (MBPS) at 2, 6, 12, and 18 month;. H5. higher maternal infant interaction scores measured using Measure of Adult and Infant Soothing and Distress Scale (MAISD) at 2, 6, 12 and 18 months.

Sample size: The sample size is 159 mother-infant dyads at 18 months.

Benefits of the Research Project: New evidence about the long-term impact of early KC provided during early painful procedures is important to the effective management of procedural pain and development in vulnerable infants. By fully integrating mothers and families as active participants, it will have direct implications regarding the improvement of outcomes of at-risk newborns, not only for their immediate physiological stability and later development, but also their families, and the health care system in general.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the original TRAKC trial (Born less than 36 6/7 weeks gestational age and were stable enough to be held in KC)
* Participants live within 100 km from hospital or are willing to routinely return to the IWK for follow-up

Exclusion criteria from the initial TRAKC trial included major congenital anomalies, receiving narcotics, or surgery.

Ages: 2 Months to 20 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Eligible parents of TRAKC infants who have provided consent will be invited back to an IWK clinic for follow-up visits at a convenient date within +/- 2 weeks of 2, 6, 12 and 18 month CA for their vaccinations as well as at 18 month corrected age for a Bayley Scales of Infant Development (BSID-III).
Sampling Method: Non-Probability Sample
Enrollment: 159 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Bayley Scales of Infant Development (BSID-III) | 18 months corrected postnatal age
  The Bayley Scales of Infant and Toddler Development (3rd edition; BSID-III) , the most widely used standardized assessment of early milestone-based development in young children, evaluates five domains related to development of infants from 1 to 42 months of age: cognitive, language, motor, adaptive behaviour, and social-emotional.

SECONDARY OUTCOMES:
Brief Infant Toddler Social Emotional Assessment (BITSEA) | 18 month corrected postnatal age
  The BITSEA is the Brief form of the Infant Toddler Social and Emotional Assessment, which covers domains of behaviour. The BITSEA is effective for children aged 12 to 36 months.
Early Childhood Behaviour Questionnaire (ECBQ) | 18 month corrected postnatal age
  The ECBQ was developed and validated to measure temperament in toddlers between 18 and 36 months of age and has shown adequate levels of reliability and validity. The 201-item parent-report questionnaire assesses 18 dimensions of temperament.
Modified Behavioral Pain Scale (MBPS) | 2, 6, 12, and 18 months
  The MBPS, a well-validated acute pain scale used to measure procedural pain, including needle related pain in infant populations, starting at 2 months. The MBPS assesses pain in terms of three observable behaviours: facial expressions, cry, and body movement.
Measure of Adult and Infant Soothing and Distress Scale (MAISD) | 2, 6, 12, and 18 months
  This is a behavioural measure developed to assess adult and infant behaviour during medical procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Marsha Campbell-Yeo, RN, NNP, PhD, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided